CLINICAL TRIAL: NCT07194070
Title: Global Prospective Hemolytic Disease of the Fetus and Newborn Registry
Brief Title: A Study on Hemolytic Disease of the Fetus and Newborn (HDFN) Through Global Registry
Acronym: GERANIUM
Status: Recruiting | Type: Observational
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: NOPRODEBF0001; NOPRODEBF0001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2025-09-11; First posted 2025-09-26 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Hemolytic Disease of the Fetus and Newborn
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant Participants at Risk for Hemolytic Disease of the Fetus and Newborn (HDFN): Pregnant participants with a risk for HDFN in their current pregnancy will be enrolled. No treatment will be provided by the sponsor as a part of this study. Only data will be collected for participants for the duration of their pregnancy and for 2 years following birth for their corresponding neonate/infant/child. Data will be collected from eligible participants at medical centers that routinely diagnose and treat pregnant participants with HDFN. Additionally, participants will be asked to complete versions of clinical outcome assessments (Patient-reported outcomes [PROs]/Observer-reported outcomes [ObsROs]) at specific times throughout follow-up. Data collection will be considered complete for eligible participants if all available data have been recorded in the electronic case report form (eCRF).
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: Standard of Care — No study treatment will be administered as part of this study. Participants will receive standard of care therapy as per local clinical practice.

SUMMARY:
The purpose of this non-interventional study is to prospectively evaluate the risk of anemia (decreased red blood cells) in fetuses (baby before birth) and neonates (baby just after birth) of pregnant participants who are at risk for hemolytic disease of the fetus and newborn (HDFN) and receiving standard of care (SoC). HDFN is a blood disease that occurs in babies before birth or just after birth when the blood types of the pregnant individual and babies are incompatible, thus resulting in fast breakdown of red blood cells (RBCs) of the fetus/baby.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant with an estimated gestational age (GA) (based on ultrasound dating) up to week 24
* History of a previous alloimmunized pregnancy that included at least one of the following: Fetal anemia diagnosed by middle cerebral artery (MCA) doppler ultrasound; Received greater than or equal to (>=) 1 intrauterine transfusion (IUT) as a result of hemolytic disease of the fetus and newborn (HDFN); Fetal hydrops; Stillbirth or fetal demise with fetal or placental pathology indicative of HDFN; Neonatal exchange transfusion due to HDFN; Neonatal simple transfusion due to HDFN; Neonatal hyperbilirubinemia due to HDFN; Positive direct antiglobulin test (DAT) in neonate
* Documented presence of maternal alloantibody based on local laboratory results during current pregnancy
* Evidence of an antigen-positive fetus corresponding to the current maternal alloantibody: Fetal antigen status confirmed by cell-free fetal DNA (cffDNA); OR Fetal antigen status confirmed by amniocentesis; OR Paternal genotype confirmed
* Pregnant participant or a legally acceptable representative has provided informed consent (per local regulations or ethics committee requirements) for the collection and use of their medical data and the medical data for their corresponding fetuses/neonates/infants/children

Exclusion Criteria:

* Participant actively participating in an interventional trial of an investigational agent
* At risk for HDFN due to ABO being the sole alloimmunization antigen in the current pregnancy (that is, ABO plus another antigen is permissible)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include pregnant participants with a risk for hemolytic disease of the fetus and newborn (HDFN) in their current pregnancy by virtue of having a previous alloimmunized pregnancy with a gestation that included fetal anemia, received intrauterine transfusion (IUT), fetal hydrops, stillbirth with fetal or placental pathology indicative of HDFN, neonatal exchange transfusion, neonatal hyperbilirubinemia due to HDFN, or positive direct antiglobulin test (DAT) in the neonate.
Sampling Method: Non-Probability Sample
Enrollment: 175 (Estimated)
Dates: Start 2025-12-17 (Actual); Primary Completion 2030-05-26 (Estimated); Study Completion 2030-09-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of Pregnancies That did not Result in Fetal Loss, Intrauterine Transfusion (IUT), Hydrops Fetalis, or Neonatal Death During the Neonatal Period | From conception through 4 weeks of age or 41 weeks PMA, whichever is later
  Percentage of pregnancies that did not result in fetal loss (due to any reason), IUT, hydrops fetalis, or neonatal death (due to any reason) during the neonatal period will be reported. Hydrops fetalis is defined as the presence of greater than or equal to (>=) 2 abnormal fluid collections in the fetus or neonate, such as ascites, pleural effusions, pericardial effusion, and generalized skin edema (skin thickness greater than [>] 5 millimeter [mm]). Post-menstrual age (PMA) is the time elapsed between the first day of the last menstrual period and birth (gestational age) plus the time elapsed after birth (chronological age).

SECONDARY OUTCOMES:
Number of Participants With Hemolytic Disease of the Fetus and Newborn (HDFN) by Severity | Through 4 weeks of age or 41 weeks PMA, whichever is later
  Number of participants in each HDFN severity index category will be reported. The severity of HDFN is defined as: 5 (fatal): fetal or neonatal death due to any reason; 4 (severe): hydrops fetalis (in fetus or newborn) or receiving IUT during pregnancy as a result of HDFN but not 5 (fatal); 3 (moderate): neonatal exchange transfusions received as a result of HDFN related hemolysis and jaundice but not 4 (severe) or 5 (fatal); 2 (mild): neonatal simple transfusions received due to HDFN after birth, with or without phototherapy, but not 3 (moderate), 4 (severe), or 5 (fatal); and 1 (minimal or none): not in 2 (mild), 3 (moderate), 4 (severe), or 5 (fatal) as described above. HDFN requiring phototherapy will be classified in this category.
Time to First Occurrence of IUT or Hydrops Fetalis | From conception to delivery date (up to maximum of 42 weeks)
  Time to first occurrence of IUT or hydrops fetalis will be reported.
Modified Neonatal Morbidity and Mortality Index (mNMMI) in Live Newborn Neonates | Through 38 weeks PMA or at discharge if earlier than 38 weeks PMA
  The mNMMI will be assessed with the following categories: fatal: neonatal death; major morbidity: any of intraventricular hemorrhage grade 3/4, seizures, hypoxic-ischemic encephalopathy, necrotizing enterocolitis stage 2/3, respiratory distress syndrome requiring mechanical ventilation, bronchopulmonary dysplasia requiring oxygen support, or persistent pulmonary hypertension; Minor morbidity: anemia requiring simple transfusion, hyperbilirubinemia requiring an exchange transfusion, hypotension requiring treatment, intraventricular hemorrhage grade 1/2, necrotizing enterocolitis stage 1, or respiratory distress syndrome not requiring mechanical ventilation; None: no major or minor morbidities described above. Hyperbilirubinemia requiring phototherapy will be classified in this category.
Number of IUTs Received During the Pregnancy | From conception to delivery date (up to maximum of 42 weeks)
  Number of IUT's received during the pregnancy will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (7):
- United States (3):
  - Riley Children s Hospital, Indianapolis, Indiana
  - University of Cincinnati, Cincinnati, Ohio
  - Baylor College of Medicine, Houston, Texas
- Interdiszip Schwerpunkt fur Hamostaseologie, Giessen, Germany
- Italy (2):
  - Mangiagalli Clinic IRCCS Ca Granda Foundation Ospedale Maggiore Policlinico, Milan
  - Fondazione Policlinico Universitario A Gemelli IRCCS, Roma
- Birmingham Women's Hospital, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No